CLINICAL TRIAL: NCT07286240
Title: A Single-arm, Multicenter Phase II Clinical Study of QL1706 Combined With Chemotherapy and Anlotinib for the Treatment of Recurrent Ovarian Cancer
Brief Title: QL1706 Combined With Chemotherapy and Anlotinib for the Treatment of Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Lipai Chen, Chief physician, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL-0ca-QIBA-3003
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Treatment of Recurrent Ovarian Cancer
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 plus chemotherapy and anlotinib regimen (Experimental)
  Interventions: Drug: QL1706 plus chemotherapy and anlotinib regimen

INTERVENTIONS:
Drug: QL1706 plus chemotherapy and anlotinib regimen — QL1706 (5 mg/kg) IV d1, q3w Pegylated liposomal doxorubicin hydrochloride (30 mg/m²) IV d1, q3w Carboplatin (AUC = 5) IV d1, q3w -OR- cisplatin (75 mg/m²) IV d1, q3w Anlotinib: 8 mg PO qd d1-14, q3w Administer for 6 cycles.

SUMMARY:
Ovarian cancer is one of the most common gynecologic malignancies, with considerable histologic heterogeneity; more than 90 % of cases are epithelial ovarian cancers. Because no reliable tools exist for early detection, approximately 70 % of patients are diagnosed at an advanced stage and have poor prognosis, and >70 % experience relapse within 3 years of initial treatment. The standard first-line strategy combines cytoreductive surgery, platinum-based chemotherapy, and maintenance with PARP inhibitors. Management of recurrent disease remains one of the most challenging problems in clinical oncology.

Bevacizumab, a recombinant humanized anti-VEGF monoclonal antibody that blocks endothelial proliferation and neovascularization, is the prototypic angiogenesis inhibitor used in ovarian cancer. However, randomized trials have demonstrated only progression-free survival (PFS) benefit, with no overall survival (OS) advantage. Pre-clinical data suggest that immunotherapy and anti-angiogenic agents can exert synergistic anti-tumor activity, yet clinical efforts combining bevacizumab with immune-checkpoint inhibitors in recurrent ovarian cancer-whether added to platinum-based chemotherapy, used as maintenance, or evaluated in chemotherapy-free regimens-have thus far been unsuccessful (except in clear-cell histology).

Anlotinib is a novel oral multi-target tyrosine-kinase inhibitor that blocks VEGFR-2/3, FGFR 1-4, PDGFR-α/β, c-KIT, and RET, thereby potently suppressing angiogenesis. Accumulating evidence indicates that anlotinib plus chemotherapy is more effective than chemotherapy alone in advanced or recurrent ovarian cancer, with a manageable safety profile, showing encouraging efficacy and tolerability.

Because conventional approaches for recurrent ovarian cancer are limited-particularly once platinum resistance develops-new therapeutic strategies are urgently needed. The best-characterized immune-checkpoint molecules are CTLA-4 and the PD-1/PD-L1 axis. Combined blockade of CTLA-4 and PD-1 has yielded impressive activity in several tumor types. Although single-agent checkpoint inhibitors produce modest response rates in recurrent ovarian cancer, preliminary data suggest that dual inhibition with anti-CTLA-4 plus anti-PD-1 antibodies may enhance therapeutic responses.QL1706 is a novel dual-target immunotherapeutic agent that has been approved for second-line monotherapy in cervical cancer.QL1706, developed by Qilu Pharmaceutical using the proprietary MabPair™ platform, is the first bispecific antibody simultaneously targeting PD-1 and CTLA-4, showing synergistic anti-tumor activity and favorable tolerability.The treatment of recurrent ovarian cancer remains a formidable challenge; therefore, proactive exploration of diverse combination regimens is essential to achieve optimal therapeutic efficacy and maximize survival benefit for patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.Capable of understanding and voluntarily signing the written Informed Consent Form (ICF); the ICF must be signed before any study-specific procedures are performed.

  2.Female, aged 18-70 years at the time of ICF signature. 3.Eastern Cooperative Oncology Group (ECOG) performance status 0-1. 4.Life expectancy ≥ 3 months. 5.Histologically confirmed epithelial ovarian cancer (including fallopian-tube and primary peritoneal carcinoma) that has recurred after standard platinum-based therapy:
  1. Platinum-sensitive relapse (recurrence ≥ 6 months after completion of the last platinum-based therapy).
  2. Platinum-resistant relapse (recurrence < 6 months after completion of the last platinum-based therapy or progression while on PARP-inhibitor maintenance).

     Note: Maintenance PARP inhibitor or bevacizumab after CR/PR to prior chemotherapy, and hormonal therapy, are not counted as additional lines of therapy.

     6.At least one measurable lesion per RECIST v1.1. Lesions previously irradiated or treated with other loco-regional therapy can serve only as non-target lesions unless clear progression is documented or tumor viability is biopsy-proven.

     7.Archived or freshly obtained tumor tissue (primary or relapse) must be available for biomarker analyses. Five unstained formalin-fixed paraffin-embedded (FFPE) slides or a tissue block are required for central PD-L1 testing (slides preferred). If re-biopsy is judged unsafe, the number of slides may be reduced after discussion with the medical monitor.

     8.Adequate organ function at screening:

     Hematology:

     Hb ≥ 90 g/L ANC ≥ 1.5 × 10⁹/L PLT ≥ 100 × 10⁹/L

     Biochemistry:

     Albumin ≥ 29 g/L ALT/AST < 3 × ULN (< 5 × ULN if liver metastases) TBIL ≤ 1.5 × ULN Creatinine ≤ 1.5 × ULN 9.Women of child-bearing potential must have a negative serum pregnancy test within 3 days before first dose. If sexually active with a non-sterilized male partner, they must use a highly effective contraceptive method from screening until 6 months after the last study-dose; rhythm or withdrawal methods are not acceptable.

     10.The need for additional cytoreductive surgery is at the investigator's discretion.

     Exclusion Criteria:
* 1.Non-epithelial ovarian malignancies (e.g., carcinosarcoma, sex-cord stromal tumors).

  2.Central-nervous-system metastases or meningeal carcinomatosis. 3.Pleural, pericardial, or ascitic effusions requiring repeat drainage > once per month.

  4.Active malignancy within 3 years before first dose, except locally curable cancers deemed cured (e.g., squamous- or basal-cell skin cancer, superficial bladder cancer, ductal carcinoma in situ of breast).

  5.Prior systemic anti-cancer therapy within 3 weeks (chemotherapy, bevacizumab/biosimilars, TKI, PARP inhibitor); palliative radiotherapy or immunomodulators (e.g., thymosin, interferon, IL-2) or cancer-treating Chinese patent medicines (e.g., Aidi injection) within 2 weeks; hormonal agents (e.g., tamoxifen, letrozole) within 1 week.

  6.Previous immune-checkpoint inhibitors (anti-PD-1, anti-PD-L1, anti-CTLA-4, etc.) or agonists of immune co-stimulatory molecules (ICOS, CD40, CD137, GITR, OX40, etc.).

  7.Major surgery, open biopsy, or significant trauma within 4 weeks; elective major surgery planned during study.

  8.Active or likely recurrent autoimmune disease (exceptions: vitiligo, alopecia, psoriasis/eczema not requiring systemic therapy; hypothyroidism from autoimmune thyroiditis on stable replacement; type 1 diabetes on stable insulin).

  9.Systemic corticosteroids > 10 mg/day prednisone equivalent or other immunosuppressants within 14 days (inhaled, ophthalmic, or topical steroids ≤ 10 mg/day permitted).

  10.Live vaccine within 4 weeks. 11.Primary or secondary immunodeficiency, including positive HIV antibody. 12.Prior solid-organ or allogeneic hematopoietic-stem-cell transplant. 13.History of interstitial lung disease or non-infectious pneumonitis. 14.Severe infection within 4 weeks (complicated infection requiring hospitalization, sepsis, severe pneumonia).

  15.Active infection requiring systemic therapy (including active TB or active syphilis) or systemic antibiotics/antivirals/antifungals within 2 weeks (except suppressive anti-HBV therapy).

  16.Active hepatitis B (HBsAg-positive with HBV DNA > 1000 IU/mL); active hepatitis C. Inactive HBV carriers with HBV DNA ≤ 1000 IU/mL are eligible. Subjects with cured HCV (HCV Ab-positive and HCV RNA-negative) are eligible.

  17.Inflammatory bowel disease (Crohn's, ulcerative colitis), active diverticulitis, clinical bowel obstruction, or need for parenteral hydration/nutrition or nasogastric tube.

  18.Significant cardiovascular/cerebrovascular disease:
  1. MI, unstable angina, pulmonary embolism, aortic dissection, DVT, arterial thrombo-embolism within 6 months
  2. NYHA class ≥ II heart failure
  3. Serious arrhythmia requiring chronic therapy (stable-rate asymptomatic atrial fibrillation allowed)
  4. CVA within 6 months
  5. LVEF < 50 %
  6. Prior myocarditis/cardiomyopathy; uncontrolled hypertension (> 150/100 mmHg) or hypertensive crisis/encephalopathy 19.Peripheral neuropathy ≥ grade 2 (NCI CTCAE v5.0). 20.Unresolved toxicity > grade 1 from prior anti-cancer therapy (except alopecia).

     21.Severe hypersensitivity to any monoclonal antibody. 22.Pregnancy or lactation. 23.Any condition that, in the investigator's opinion, would compromise safety, interfere with study evaluations, or confound results (e.g., severe concomitant disease or psychiatric disorder).

     24.Known hypersensitivity to any study drug or excipient. 25.Prior gastrointestinal perforation, intra-abdominal abscess, or bowel obstruction within 3 months or radiologic/clinical evidence of obstruction.

     26.Hypertension inadequately controlled on medication (systolic ≥ 140 mmHg or diastolic ≥ 90 mmHg).

     27.Coagulopathy (INR > 2.0 or PT > 16 s), bleeding diathesis, or thrombolytic/anticoagulant therapy (prophylactic low-dose aspirin or LMWH allowed).

     28.Clinically significant bleeding or bleeding tendency within 3 months (e.g., GI bleeding, hemorrhagic gastritis, vasculitis).

     29.Arterial or venous thrombosis within 6 months (CVA, TIA, intracranial bleed, DVT, PE); superficial vein thrombosis may be allowed at investigator's discretion.

     30.Hereditary or acquired bleeding/thrombotic disorders (e.g., hemophilia, coagulation defects, thrombocytopenia).

     31.Active ulcer, non-healing wound, or fracture. 32.Urine protein ≥ ++ confirmed by 24-h urine protein > 1.0 g. 33.Prior palliative radiotherapy to > 5 % of bone-marrow area within 4 weeks. 34.Strong CYP3A4 inducers within 2 weeks or strong CYP3A4 inhibitors within 1 week.

     35.Prior treatment with anlotinib or other small-molecule multi-target TKIs.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The ratio of patients who are evaluated as CR or PR
PFS | 2 years
  PFS: defined as the time from the date of first dose to the first documented progressive disease (PD) or death from any cause, whichever occurs first, within the tumor-assessment follow-up period.

SECONDARY OUTCOMES:
DCR | 2 years
  DCR: the proportion of patients with best overall response of complete response (CR), partial response (PR), or stable disease (SD) for ≥4 weeks.
OS | 2 years
  OS: defined as the time from the date of first dose to death from any cause (for patients lost to follow-up before death, the date of last known contact is conventionally used as the date of death).
DOR | 2 years
  DOR: In patients who achieve an objective response, DOR is defined as the time from the first documented complete response (CR) or partial response (PR) (whichever occurs first) to the date of progressive disease (PD) or death from any cause (whichever occurs first).
TTR | 2 years
  TTR (Time to Response): For patients who achieve an objective response, TTR is defined as the time from the date of first dose to the first documented complete response (CR) or partial response (PR), whichever occurs first.
CA125 response | 2 years
  CA125 response: assessed according to the GCIG (Gynecologic Cancer InterGroup) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Lipai Chen, Guangzhou, Guangdong, China